CLINICAL TRIAL: NCT06323798
Title: Diffusion Weighted MRI Enables Differential Diagnosis Between Pyocele and Mucocele
Status: Not yet recruiting | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2024PI035
Record Dates: First submitted 2024-03-15; First posted 2024-03-21 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Pyocele; Sinus
Keywords: sinus, pyocele, mri
MeSH Terms: conditions — Fistula

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- cases: patients with a paranasal sinus mri and a confirmed pyocele at bacteriologic sample reviewed in the medical file
  Interventions: Diagnostic Test: MRI
- controls: patients with a paranasal sinus mri and a confirmed simple retention mucus at bacteriologic sample reviewed in the medical file
  Interventions: Diagnostic Test: MRI

INTERVENTIONS:
Diagnostic Test: MRI — Standard paranasal sinus MRI

SUMMARY:
Diffusion MRI should allow for differentation of pus and simple retention in the paranasal sinuses, but this remained to be determined

DETAILED DESCRIPTION:
On the basis of the apparent diffusion coefficient, the content of a para nasal sinus could be defined as simple mucus or pus. This differentiation is very important for the clinician for prompt treatment. The aim of this study is to retrospectively measure this coefficient and to correlate it to clinica data.

ELIGIBILITY:
Inclusion Criteria:

* paranasal sinus MRI with a diffusion weighted sequence

Exclusion Criteria:

* no clinical examination available
* no bateriologic sample available

Ages: 18 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients with paranasal MRI
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-04-28 (Estimated); Primary Completion 2024-07-28 (Estimated); Study Completion 2024-12-28 (Estimated)

PRIMARY OUTCOMES:
apparent diffusion coefficient | 5 years
  apparent diffusion coefficient on a diffusion weighted MRI sequence

CONTACTS AND LOCATIONS:
Overall Officials: romain gillet, md, Principal Investigator — CHRU de Nancy

IPD SHARING:
Plan to Share IPD: No
MRI is the proprety of the patient

REFERENCES:
- [Background] Radulesco T, Scemama U, Mancini J, Moulin G, Dessi P, Michel J, Varoquaux A. Role of diffusion-weighted imaging in the discrimination of purulent intrasinusal content: A retrospective study. Clin Otolaryngol. 2019 Sep;44(5):762-769. doi: 10.1111/coa.13388. Epub 2019 Jul 23. PMID 31169984